CLINICAL TRIAL: NCT03657745
Title: An Observational Trial of Alzheimer's Disease Treatment With Combination of 40Hz Light and Cognitive Therapy
Brief Title: Alzheimer's Disease Treatment With Combination of 40Hz Light and Cognitive Therapy
Acronym: AlzLife
Status: Recruiting | Type: Observational
Sponsor: Alzheimer's Light LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: AlzLife001
Record Dates: First submitted 2018-08-16; First posted 2018-09-05 (Actual); Last update posted 2024-08-01 (Actual); Status verified 2024-07

CONDITIONS: Alzheimer Disease; Mild Cognitive Impairment; Dementia; Cognition Disorders in Old Age; Cognitive Decline; Cognitive Deterioration
Keywords: Alzheimer Disease; Alzheimer's; Dementia
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction; Dementia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Participants who adhere to the protocol: All participants are encouraged to exercise with AlzLife daily for 30 minutes a day. The actual duration is to be measured through participant's interactions with ALZLIFE. Participants adhere to the protocol if they exercise with AlzLife the minimum of 1hour/week.
  Interventions: Device: Combination of 40Hz light and cognitive therapy (ALZLIFE)
- Participants who do not adhere to the protocol: All participants are encouraged to exercise with AlzLife daily for 30 minutes a day. The actual duration is to be measured through participant's interactions with ALZLIFE. Participants do not adhere to the protocol if they exercise with AlzLife less than 1hour/week.
  Interventions: Device: Combination of 40Hz light and cognitive therapy (ALZLIFE)

INTERVENTIONS:
Device: Combination of 40Hz light and cognitive therapy (ALZLIFE) — Combination of 40Hz light and cognitive therapy delivered by iPad application ALZLIFE

SUMMARY:
Electrical activity in the brain known as "gamma" brainwaves help connect and process information throughout the brain. These gamma waves are diminished in Alzheimer's disease. New research in Alzheimer's disease mouse models shows that exposure to light flickering at the rate of 40 flashes per second or 40Hz increased gamma brainwaves and led to clearing of beta amyloid plaques in the brain, a key abnormality in Alzheimer's disease. This project will test the ability of a novel iPad App (AlzLife https://www.alz.life/) that delivers light therapy at 40 Hz combined with cognitive therapy to improve cognition, function, and quality of life in Alzheimer's disease.

DETAILED DESCRIPTION:
New research suggests that exposure to a light flickering at 40Hz may promote gamma brain wave activity through the photic entrainment phenomenon. These waves have the potential to activate critical cleaning cells in the brain that could eliminate beta amyloid plaques. The most recent research on light therapy for Alzheimer's disease appeared in the journal Nature in 2017, entitled "How flashing lights and pink noise might banish Alzheimer's, improve memory and more" (the full article can be freely accessed at: https://www.nature.com/articles/d41586-018-02391-6) and in 2016, entitled "Gamma frequency entrainment attenuates amyloid load and modifies microglia" (the article abstract can be accessed at: https://www.nature.com/articles/nature20587). Researchers from MIT found that shining a strobe light into the eyes of mice with a rodent version of Alzheimer's disease encouraged protective cells to phagocytize the harmful proteins that accumulate in the brain. The perfect rate of flashes was determined to be 40 per second. Exposure to the flashing light for an hour (light therapy) led to a noticeable reduction in beta amyloid levels the next day in regions of the neocortex and hippocampus. When done every day for a week, beta amyloid levels were greatly reduced.

In addition, there is a significant body of evidence that computerized brain training (cognitive therapy) improves the memory of patients with Alzheimer's and dementia, which could help avert some symptoms of cognitive decline.

The synergistic combination of light and cognitive therapy utilized in AlzLife has the potential to improve the brain's function better than either of these therapies alone. This project will test the ability of a novel iPad App ("ALZLIFE") that delivers light therapy at 40 Hz combined with cognitive therapy to improve cognition, function, and quality of life in Alzheimer's disease.

ELIGIBILITY:
Inclusion Criteria:

* Alzheimer's disease
* Cognitive Impairment

Exclusion Criteria:

* any previously noted epileptic seizures, including febrile seizures.
* any significant disease of the eye, such as macular degeneration. Since the 40Hz light therapy is delivered via eye stimulation, healthy eyes are required.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Alzheimer's disease and Cognitive Impairment
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
In-app cognitive test | through study completion, an average of 1 year
  The cognitive therapy delivered by ALZLIFE consist of cognitive games: Sudoku, Tic-Tac-Toe, Analog clock comparison, etc. The changes in performance score in these cognitive games are used to calculate the participant's Cognitive Index.
  Cognitive Index maximum score = 100. The lower score indicates worse performance.

SECONDARY OUTCOMES:
Alzheimer's Disease Cooperative Study-activities of daily living (ADCS-ADL) | through study completion, an average of 1 year
  The ADCS-ADL assesses the competence of patients with Alzheimer's Disease (AD) in basic and instrumental activities of daily living (ADLs). ADCS-ADL is assessed by an in-app evaluation completed by a caregiver every month. All responses relate to the 4 weeks prior to the time of rating. The six basic ADL items each take an ADL (e.g., eating) and provide descriptions of level of competence, with the rater selecting the most appropriate option (e.g., ate without physical help and used a knife; used a fork or spoon but not a knife; used fingers to eat; was usually fed by someone else). ADCS-ADL maximum score = 30. The lower score indicates worse outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Andrey Vyshedskiy, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Iaccarino HF, Singer AC, Martorell AJ, Rudenko A, Gao F, Gillingham TZ, Mathys H, Seo J, Kritskiy O, Abdurrob F, Adaikkan C, Canter RG, Rueda R, Brown EN, Boyden ES, Tsai LH. Gamma frequency entrainment attenuates amyloid load and modifies microglia. Nature. 2016 Dec 7;540(7632):230-235. doi: 10.1038/nature20587. PMID 27929004
- [Background] Thomson H. How flashing lights and pink noise might banish Alzheimer's, improve memory and more. Nature. 2018 Mar 1;555(7694):20-22. doi: 10.1038/d41586-018-02391-6. No abstract available. PMID 29493598
- [Background] Martorell AJ, Paulson AL, Suk HJ, Abdurrob F, Drummond GT, Guan W, Young JZ, Kim DN, Kritskiy O, Barker SJ, Mangena V, Prince SM, Brown EN, Chung K, Boyden ES, Singer AC, Tsai LH. Multi-sensory Gamma Stimulation Ameliorates Alzheimer's-Associated Pathology and Improves Cognition. Cell. 2019 Apr 4;177(2):256-271.e22. doi: 10.1016/j.cell.2019.02.014. Epub 2019 Mar 14. PMID 30879788
- See also: ALZLIFE website — https://www.alz.life/
- See also: ALZLIFE application in the App Store — https://itunes.apple.com/us/app/alzheimers-light-therapy/id1327175926?mt=8